CLINICAL TRIAL: NCT07109414
Title: Randomized Phase 2/3 Trial of NP-G2-044 (Prilukae) Combined With PLD for Treatment of Platinum-Resistant Ovarian Cancer (ULTIMUS-1)
Brief Title: Trial of NP-G2-044 (Prilukae) Combined With PLD for Treatment of Platinum-Resistant Ovarian Cancer (ULTIMUS-1)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novita Pharmaceuticals, Inc. (Industry)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP-G2-044-P3-01; GOG-3121 (Other: Gynecologic Oncology Group)
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Platinum-resistant Ovarian Cancer
Keywords: Dose escalation; Dose optimization; Small-molecule fascin inhibitor; Advanced or metastatic ovarian cancer; Randomized Phase 3
MeSH Terms: conditions — Ovarian Neoplasms | interventions — NP-G2-044; 1-dodecylpyridoxal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A1 (Dose escalation):NP-G2-044 Monotherapy (Experimental): Participants will receive multiple doses of NP-G2-044 in tablet form orally as a monotherapy twice a daily.
  Interventions: Drug: NP-G2-044
- Part A2 (Dose escalation): NP-G2-044+PLD combination therapy (Experimental): Participants will receive multiple doses of NP-G2-044 (once daily [QD] or BID) in tablet form orally plus a single dose of PLD as an infusion via intravenous route once in every 28 days. The recommended monotherapy doses of NP-G2-044 are determined from the results of Part A1.
  Interventions: Drug: NP-G2-044; Drug: PLD
- Part B (Dose optimization): NP-G2-044+PLD combination dose level 1 (Experimental): Participants will receive daily dose of NP-G2-044 in tablet form orally plus a single dose of PLD as an infusion via intravenous route once in every 28 days.
  Interventions: Drug: NP-G2-044; Drug: PLD
- Part B (Dose optimization): NP-G2-044+PLD combination dose level 2 (Experimental): Participants will receive daily dose of NP-G2-044 in tablet form orally plus a single dose of PLD as an infusion via intravenous route once in every 28 days.
  Interventions: Drug: NP-G2-044; Drug: PLD
- Part B (Dose optimization) :PLD (Active Comparator): Participants will receive a single dose of PLD as an infusion via intravenous route alone once in every 28 days.
  Interventions: Drug: PLD
- Part C (Phase 3): NP-G2-044+PLD (Experimental): Participants will receive daily dose of NP-G2-044 in tablet form orally plus a single dose of PLD as an infusion via intravenous route once in every 28 days.
  Interventions: Drug: NP-G2-044; Drug: PLD
- Part C (Phase 3): PLD (Active Comparator): Participants will receive a single dose of PLD as an infusion via intravenous route once in every 28 days.
  Interventions: Drug: PLD

INTERVENTIONS:
Drug: NP-G2-044 — NP-G2-044 will be provided as a tablet via oral route of administration in the study.
  Other Names: Prilukae
  Arms: Part A1 (Dose escalation):NP-G2-044 Monotherapy; Part A2 (Dose escalation): NP-G2-044+PLD combination therapy; Part B (Dose optimization): NP-G2-044+PLD combination dose level 1; Part B (Dose optimization): NP-G2-044+PLD combination dose level 2; Part C (Phase 3): NP-G2-044+PLD
Drug: PLD — PLD will be provided as an infusion via intravenous route of administration in the study.
  Arms: Part A2 (Dose escalation): NP-G2-044+PLD combination therapy; Part B (Dose optimization) :PLD; Part B (Dose optimization): NP-G2-044+PLD combination dose level 1; Part B (Dose optimization): NP-G2-044+PLD combination dose level 2; Part C (Phase 3): NP-G2-044+PLD; Part C (Phase 3): PLD

SUMMARY:
The purpose of the study is to identify the optimal dose level of NP-G2-044 in combination with standard of care (SOC) pegylated liposomal doxorubicin (PLD), and to compare the efficacy and safety of NP-G2-044+PLD vs. PLD alone in participants with platinum-resistant ovarian cancer (PROC).

DETAILED DESCRIPTION:
This is an open-label, Phase 2/3, multicenter, randomized study of NP-G2-044 in combination with PLD vs. PLD alone in participants with PROC. The Phase 2 component of the study includes a safety lead-in dose escalation of NP-G2-044 monotherapy with twice daily (BID) dosing and a dose escalation phase for NP-G2-044+PLD followed by a randomized dose optimization phase of NP-G2-044+PLD compared with PLD. In the Phase 3 component of the study, participants will be randomized to treatment with NP-G2-044+PLD, at the dose selected from the dose optimization phase, or to PLD alone. Randomized participants will be stratified according to the number of prior lines of therapy, number of prior PLD therapy lines, and region of the world. The study population is women at least 18 years of age with confirmed ovarian high grade serous carcinoma, an Eastern Cooperative Oncology Group (ECOG) status of 0-1, and whose cancer is resistant to platinum-based therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have confirmed ovarian high-grade serous carcinoma (histologically or cytologically)

  1. Participants should have platinum resistance
  2. No PLD use after developing platinum resistance
  3. Participants must have had bevacizumab in a prior treatment line or must have been ineligible for bevacizumab therapy.
* ECOG status 0-1
* Measurable disease per RECIST v1.1 as assessed by local site Investigator/radiologists in the Dose Escalation phase, and assessed by BICR in the Dose Optimization phase and Phase 3; lesions situated in previous irradiated areas are considered measurable if progression has been demonstrated in such lesions
* Left ventricular ejection fraction > 50%
* Participants with adequate hematologic function based on following

  1. Absolute neutrophil count ≥ 1.5 × 109/L
  2. Platelet count ≥ 100 × 109/L
  3. Hemoglobin ≥ 9.0 g/dL
  4. Albumin ≥ 3.0 g/dL
* Adequate coagulation parameters based on the following:

  1. Prothrombin time-internationalization normal rate (INR)/partial thromboplastin time < 1.5 × upper limit of normal (ULN)
  2. Partial thromboplastin time or activated partial thromboplastin time < 1.25 × ULN
* Participants must have adequate hepatic and renal function. For hepatic function, total bilirubin should be less than 1.5 times the ULN. For renal function, serum creatinine clearance must be at least 45 mL/min.
* Participants of childbearing potential (defined as sexually mature women who have not undergone surgical sterilization or been postmenopausal for at least 12 months if over 55 years of age) must have a negative pregnancy test within 72 hours before starting treatment. These participants must use highly effective contraception or abstain from heterosexual activity from screening through 120 days after the last dose of study medication.

Exclusion Criteria:

* Primary platinum-refractory (recurrence within 120 days of first-line platinum-containing therapy or during first-line platinum-containing therapy).
* Recurrence greater than 183 days from the penultimate platinum (platinum-sensitive recurrent ovarian cancer).
* Uncontrolled malignant pleural effusions and/or ascites as defined by a prior needle drainage within 60 days of first dose.
* Major surgery within 4 weeks prior to Screening.
* Prior radiotherapy within 4 weeks of start of study treatment.

  1. Participants must have recovered from all radiation-related toxicities, not require corticosteroids for their radiation therapy, and have no history of radiation pneumonitis.
  2. A 1-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
* Anticancer therapy, such as chemotherapy, immunotherapy, hormonal therapy, targeted therapy, or investigational agents prior to administration of the first dose of study treatment.
* Active CNS metastases; participants with leptomeningeal metastases are not eligible.
* Primary CNS malignancy.
* Severe gastrointestinal conditions such as existing bowel obstruction defined as air fluid levels in the small bowel and/or intolerance to oral medications, clinical or radiological evidence of bowel obstruction within 8 weeks prior to study entry requiring hospitalization, current use of nasogastric tube decompression, inability to tolerate solid feedings or vomiting more than once a day.
* Liver metastases involving > 60% of liver parenchyma.
* Known active infection with Human immunodeficiency virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C virus (HCV)
* Requiring immunosuppressive therapy
* Evidence of ongoing systemic bacterial, fungal, or viral infections at Screening
* Received a live vaccine within 6 weeks of first dose of study drug.
* Received a Coronavirus disease-2019 (COVID-19) vaccine less than 1 week prior to dosing (Cycle 1/Day 1) and/or during the study received a COVID-19 vaccine or booster less than 3 weeks ahead of a tumor assessment.
* Baseline QT interval corrected with Fridericia's method (i.e., QTcF) > 470 ms.
* Female participants who are pregnant or breastfeeding.
* Concurrent active malignancy.
* History of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis which required steroid treatment.
* History of stroke, unstable angina, myocardial infarction, congestive heart failure (NYHA classification III or IV), clinically significant left ventricular hypertrophy or ventricular arrhythmia requiring medication or mechanical control within the last 6 months prior to Screening.
* Participants with increased baseline risk of Torsades de Pointe due to:

  1. Electrolyte imbalance at screening (clinically significant hypokalemia, hypomagnesemia or hypocalcemia per Investigator's determination)
  2. Known congenital long QT syndrome (LTQS)
  3. Bradycardia (heart rate < 50 beats per minute)
* Unstable or severe uncontrolled medical condition like unstable cardiac function, unstable pulmonary condition including pneumonitis and/or interstitial lung disease, uncontrolled diabetes or any important medical illness or abnormal laboratory findings
* Grade 3 or 4 toxicity due to PLD in prior treatment.
* Grade 2 or greater neuropathy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 380 (Estimated)
Dates: Start 2025-12-29 (Actual); Primary Completion 2028-10-25 (Estimated); Study Completion 2029-10-24 (Estimated)

PRIMARY OUTCOMES:
Part A (Dose escalation): Number of participants with adverse events (AEs) | From first dose until Safety Follow-up (30 days ±7 days after last dose of NP-G2-044) Approximately 2 years
  The safety and tolerability of NP-G2-044 monotherapy with BID dosing and in combination with PLD will be evaluated
Part A (Dose escalation): Number of participants with Dose Limiting Toxicities (DLTs) | Up to 28 days
  The safety and tolerability of NP-G2-044 monotherapy with BID dosing and in combination with PLD and to determine the recommended Phase 2 dose (RP2D) of NP-G2-044 when combined with PLD will be determined
Part B (Dose Optimization): Number of participants with AEs | From Day 1 until Safety Follow-up (30 days ±7 days after last dose of NP-G2-044) Approximately 2 years
  The safety and tolerability of the treatment groups will be compared.
Part B (Dose Optimization): Overall response rate (ORR) | From randomization until disease progression, death, or withdrawal of consent, whichever occurs first (Approximately 2 years)
  The optimal dose of NP-G2-044 combined with PLD will be evaluated. The ORR is defined as the proportion of participants with complete response (CR) or partial response (PR).
Part B (Dose Optimization): Progression free survival (PFS) | From randomization until disease progression, death, or withdrawal of consent, whichever occurs first (Approximately 2 years)
  The optimal dose of NP-G2-044 combined with PLD will be evaluated. The PFS is defined as time from randomization until adequately documented disease progression based on blinded independent committee review (BICR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or death, whichever occurs first.
Part C (Phase 3): Progression free survival (PFS) | From randomization until disease progression, death, or withdrawal of consent, whichever occurs first (Approximately 3 years
  The efficacy of NP-G2-044 when combined with PLD vs. PLD alone will be compared. The PFS is defined as time from randomization until adequately documented disease progression based on BICR per RECIST v1.1 or death, whichever occurs first.

SECONDARY OUTCOMES:
Part A (Dose Escalation) and Part C (Phase 3): Overall response rate (ORR) | From randomization until disease progression, death, or withdrawal of consent, whichever occurs first (For Part A: Approximately 2 years; Part C: Approximately 3 years)
  The initial efficacy of NP-G2-044 in combination with PLD will be evaluated. The ORR is defined as the proportion of participants with CR or PR.
Part A (Dose Escalation): Progression free survival (PFS) | From randomization until disease progression, death, or withdrawal of consent, whichever occurs first (For Part A: Approximately 2 years; Part C: Approximately 3 years)
  The initial efficacy of NP-G2-044 in combination with PLD will be evaluated. The PFS is defined as time from start of treatment until adequately documented disease progression based on local assessment of imaging studies, or death, whichever occurs first.
Part A (Dose Escalation), Part B (Dose optimization) and Part C (Phase 3): Gynecologic Cancer Intergroup Cancer antigen-125 (GCIG CA-125) criteria for response | From Screening to survival follow-up (until progression, death, or withdrawal of consent) (For Part A and B: Approximately 2 years; Part C: Approximately 3 years)
  The initial efficacy of NP-G2-044 in combination with PLD will be evaluated. A response according to CA-125 has occurred if there is at least a 50% reduction in CA-125 levels from a pretreatment sample. The response must be confirmed and maintained for at least 28 days. Participants can be evaluated according to CA-125 only if they have a pretreatment sample that is at least twice the upper limit of normal and within 2 weeks prior to starting treatment. The date when the CA-125 level is first reduced by 50% is the date of the CA-125 response. To calculate CA-125 responses accurately, the following rules apply: 1) Intervening samples and the 28-day confirmatory sample must be less than or equal to (within an assay variability of 10%) the previous sample. 2) Variations within the normal range of CA-125 levels will not interfere with the response definition.
Part A (Dose Escalation), Part B (Dose optimization) and Part C (Phase 3): Overall survival (OS) | From randomization until death For Part A and B: Approximately 2 years; Part C: Approximately 3 years)
  The initial efficacy of NP-G2-044 in combination with PLD will be evaluated. The OS is defined as time from start of treatment until death.
Part A (Dose Escalation), Part B (Dose optimization) and Part C (Phase 3): Disease control rate (DCR) | From randomization until disease progression, death, or withdrawal of consent, whichever occurs first (For Part A and B: Approximately 2 years; Part C: Approximately 3 years)
  The initial efficacy of NP-G2-044 in combination with PLD will be evaluated. The DCR is defined as the proportion of participants with confirmed CR, PR or stable disease (SD).
Part A (Dose Escalation), Part B (Dose optimization) and Part C (Phase 3): Duration of response (DOR) | From randomization until disease progression, death, or withdrawal of consent, whichever occurs first (For Part A and B: Approximately 2 years; Part C: Approximately 3 years)
  The initial efficacy of NP-G2-044 in combination with PLD will be evaluated. The DoR is defined as the time from first CR or PR to disease progression or death in participants who achieve CR or PR.
Part A (Dose Escalation), Part B (Dose optimization) and Part C (Phase 3): Metastasis-free interval (MFI) | From treatment initiation to confirmed occurrence of new metastasis (For Part A and B: Approximately 2 years; Part C: Approximately 3 years)
  The initial efficacy of NP-G2-044 in combination with PLD will be evaluated. The MFI is defined as the time from start of treatment to confirmed occurrence of new metastasis.
Part A (Dose Escalation) and Part C (Phase 3): Number of participants with AEs | From Day 1 until Safety Follow-up (30 days ±7 days after last dose of NP-G2-044) For Part A and B: Approximately 2 years; Part C: Approximately 3 years)
  The safety and the tolerability of the treatment groups will be compared.
Part A (Dose Escalation), Part B (Dose optimization) and Part C (Phase 3): Participant reported outcomes based on European Organization for the Research and Treatment of Cancer Core Quality of Life Questionnaire-Ovarian Cancer Module 28 (EORTC QLQ-OV28) | At screening, every 3 cycles starting Cycle 1 Day 1 (each Cyle is 28 days) For Part A and B: (Approximately 2 years; Part C: Approximately 3 years)
  The treatment groups for participant reported Quality of life (QoL) will be compared. The EORTC QLQ-OV28 will evaluate the QoL with respect to ovarian cancer. The EORTC QLQ-OV28 is specific for ovarian cancer and consists of 28 items. Each scale was scored from 0 to 100 with higher scores on the symptom scales indicating greater symptom burden.
Part A (Dose Escalation), Part B (Dose optimization) and Part C (Phase 3): Participant reported outcomes based on European Quality of Life -5 Dimensions -5 Levels (EuroQol EQ-5D-5L) | At screening, every 3 cycles starting Cycle 1 Day 1 (each Cyle is 28 days) (For Part A and B: Approximately 2 years; Part C: Approximately 3 years)
  The treatment groups for participant reported QoL will be compared. The EQ-5D-5L questionnaire assess health outcome from a wide variety of interventions on a common scale. It is comprised of 5 dimensions where each dimension has 5 levels. A higher score represents a worse outcome.
Part A (Dose Escalation), Part B (Dose optimization) and Part C (Phase 3): Participant reported outcomes based on Functional Assessment of Cancer Therapy Ovarian Symptom Index (FOSI) | At screening, every 3 cycles starting Cycle 1 Day 1 (each Cyle is 28 days) (For Part A and B: Approximately 2 years; Part C: Approximately 3 years)
  The treatment groups for participant reported QoL will be compared. The FOSI 8-item questionnaire measures response to treatment based on symptom assessment. The FOSI total score ranges from 0 (severely symptomatic) to 32 (asymptomatic).
Part A (Dose Escalation) and Part B (Dose optimization): Terminal half-life (T1/2) of NP-G2-044 and PLD | From Day 1 to End of treatment (Approximately 2 years)
  The T1/2 of NP-G2-044 as a monotherapy with BID dosing and NP-G2-044 and PLD as combination therapy will be evaluated.
Part A (Dose Escalation) and Part B (Dose optimization): Time to maximum plasma concentration (Tmax) of NP-G2-044 and PLD | From Day 1 to End of treatment (Approximately 2 years)
  The Tmax of NP-G2-044 as a monotherapy with BID dosing and NP-G2-044 and PLD as combination therapy will be evaluated.
Part A (Dose Escalation) and Part B (Dose optimization): Maximum plasma concentration (Cmax) of NP-G2-044 and PLD | From Day 1 to End of treatment (Approximately 2 years)
  The Cmax of NP-G2-044 as a monotherapy with BID dosing and NP-G2-044 and PLD as combination therapy will be evaluated.
Part A (Dose Escalation) and Part B (Dose optimization): Area under the plasma concentration-time curve (AUC) of NP-G2-044 and PLD | From Day 1 to End of treatment (Approximately 2 years)
  The AUC of NP-G2-044 as a monotherapy with BID dosing and NP-G2-044 and PLD as combination therapy will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Jillian Zhang, PhD, Study Director — Novita Pharmaceuticals, Inc.; Lisa Barroilhet, MD, Principal Investigator — University of Wisconsin, Madison
Locations (5):
- United States (5):
  - HonorHealth Cancer Care, Phoenix, Arizona
  - Trials365, Shreveport, Louisiana
  - University of Pennsylvania Health System, Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Utah Cancer Specialists, Salt Lake City, Utah
  - University Of Wisconsin Carbone Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No